CLINICAL TRIAL: NCT02010814
Title: Metabolic and Endocrinological Characterization of a Prospective Cohort of Women With PCOS
Brief Title: Characterization of a Prospective Cohort of Women With PCOS
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Andersen, DMSci, Odense University Hospital
Other Study IDs: BIO; PCOS Biobank (Registry Identifier: PCOS Biobank)
Record Dates: First submitted 2013-11-21; First posted 2013-12-13 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; Inflammation; Body Composition
MeSH Terms: conditions — Polycystic Ovary Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PCOS: Women fulfilling at least two of the three Rotterdam criteria for PCOS, including
  * Irregular menstrual cycle
  * Clinical/biochemical hyperandrogenemia
  * Polycystic ovaries

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder in premenopausal women. PCOS is characterized by increase levels of testosterone, unwanted hair growth, adiposity, irregular menstrual cycle, and infertility. PCOS is associated with diabetes mellitus and cardiovascular diseases. Women with PCOS are reported to have increased levels of stress hormones, which may be associated with decreased quality of life. Increased testosterone levels in women may decrease the risk of osteoporosis. The aim of the present study is to measure levels of stress hormones in urine and describe quality of life using questionnaires. In addition we aim to characterize body composition and bone architecture using DXA and ExtremeCT.

As part of the project, a Biobank with fasting blood samples from participants is established.

ELIGIBILITY:
Inclusion Criteria:

* PCOS

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with PCOS, diagnosed by the Rotterdam criteria which include at least two of the following:
  * irregular mestrual cycle
  * polycystic ovaries
  * biochemical/clinical hyperandrogenemia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
bone mass density (BMD) | baseline
  BMD measured by DXA scans and ExtremeCT scans.

SECONDARY OUTCOMES:
Stress hormones | Baseline
  Measurement of cortisol and steroid metabolites in 24 hour urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Glintborg, MD PhD, Principal Investigator — Department of Endocrinology, Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Denmark